CLINICAL TRIAL: NCT00173485
Title: The Study of Infection and Cell Inflammation in Peritoneal Dialysate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700636
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2005-06

CONDITIONS: Peritonitis; Kidney Failure
Keywords: peritonitis, peritoneal dialysis, dialysate
MeSH Terms: conditions — Peritonitis; Renal Insufficiency

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
A progressive decline of plasma triggering receptor expressed on myeloid cells-1 (TREM-1) concentration indicates a favorable clinical evolution during the recovery phase of sepsis. The expression of TREM-1 in dialysate of peritoneal dialysis patients was not yet documented. We will collect the dialysate of peritonitis in peritoenal dialysis patients and analyze the time serial change.

DETAILED DESCRIPTION:
The triggering receptor expressed on myeloid cells-1 (TREM-1) is a member of the immunoglobulin superfamily, and its expression is upregulated on phagocytic cells in the presence of bacteria or fungi (1). Several experiments by Bouchon and colleagues showed that TREM-1 mediates the acute inflammatory response to microbial products. Human tissues infected with bacteria are infiltrated with neutrophils and macrophages that express high levels of TREM-1. Conversely, TREM-1 is only weakly expressed in samples from patients with noninfectious inflammatory disorders. In addition, TREM-1 is shed from the membrane of activated phagocytes and can be found in a soluble form in body fluids. The presence of a soluble form of TREM-1 in samples of bronchoalveolar lavage fluid from mechanically ventilated patients has been shown to be a good indicator of infectious pneumonia. During sepsis, a progressive decline of plasma sTREM-1 concentration indicates a favorable clinical evolution during the recovery phase of sepsis. In addition, baseline sTREM-1 level may prove useful in predicting outcome of septic patients. We will collect the dialysate of peritonitis in peritoneal dialysis patients and analyze the time serials change.

ELIGIBILITY:
Inclusion Criteria:

peritoneal dialysis patients, dialysis period for more than 3 months.

Exclusion Criteria:

age younger than 18 years old, Pregnant or lactating women. (Pre-menopause women, capable of bearing children will undergo pregnancy test)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-06; Study Completion 2009-06

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, MD, PhD, Study Chair — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Bouchon A, Dietrich J, Colonna M. Cutting edge: inflammatory responses can be triggered by TREM-1, a novel receptor expressed on neutrophils and monocytes. J Immunol. 2000 May 15;164(10):4991-5. doi: 10.4049/jimmunol.164.10.4991. PMID 10799849
- [Background] Bouchon A, Facchetti F, Weigand MA, Colonna M. TREM-1 amplifies inflammation and is a crucial mediator of septic shock. Nature. 2001 Apr 26;410(6832):1103-7. doi: 10.1038/35074114. PMID 11323674
- [Background] Gibot S, Cravoisy A, Levy B, Bene MC, Faure G, Bollaert PE. Soluble triggering receptor expressed on myeloid cells and the diagnosis of pneumonia. N Engl J Med. 2004 Jan 29;350(5):451-8. doi: 10.1056/NEJMoa031544. PMID 14749453